CLINICAL TRIAL: NCT04773015
Title: A Post-Authorisation Safety Study to Evaluate the Effectiveness of VIZAMYL™ Reader Training in Europe
Brief Title: A Study to Evaluate the Effectiveness of VIZAMYL™ Reader Training Programme in Europe
Status: Completed | Type: Observational
Sponsor: GE Healthcare (Industry)
Collaborators: ICON plc (Industry)
Responsible Party: Sponsor
Other Study IDs: GE-067-027
Record Dates: First submitted 2021-02-23; First posted 2021-02-26 (Actual); Results first posted 2024-10-10 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Cognitive Impairment
Keywords: Vizamyl; flutemetamol; Alzheimer's disease; cognitive impairment; dementia
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease; Dementia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a study to determine the effectiveness of the VIZAMYL™ reader training programme in clinical practice in Europe

DETAILED DESCRIPTION:
This study is a combination of Prospective and Retrospective models.

ELIGIBILITY:
Inclusion Criteria:

* The subject is an adult (aged 18 years or older) of any race or gender and has been referred for a VIZAMYL™ PET brain scan as part of the assessment of his/her cognitive impairment.
* The VIZAMYL™ scan was ordered as part of the clinical care of the subject and is not exclusively for a clinical trial.
* If informed consent is required by the local IEC, the subject, or his/her legally authorised representative, is willing and able to sign consent for use of their de-identified VIZAMYL™ PET images and associated anatomic images (brain CT and/or MRI) used in the interpretation of the VIZAMYL™ images as well as de-identified demographic information.

Exclusion Criteria:

* If informed consent is required by the local IEC, the subject (or representative) is not willing to consent to their de-identified images and other data being used in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: tertiary referral
Sampling Method: Non-Probability Sample
Enrollment: 227 (Actual)
Dates: Start 2018-12-11 (Actual); Primary Completion 2021-12-07 (Actual); Study Completion 2021-12-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Sherwin, MD, PhD, Study Director — GE Healthcare
Locations (10):
- Austria (2):
  - Kepler Universittsklinikum Neuromed Campus, Linz, Wagner-Jauregg-Weg
  - Landeskrankenhaus Vocklabruck, Vöcklabruck
- Helsinki University Central Hospital, Helsinki, Finland
- Italy (3):
  - Ospedal Mons Dimicolli - Barletta, Barletta
  - U.O. Medicina Nucleare- ASSST Spedali Civili P.O. di Brescia, Brescia
  - Azienda Ospedaliero Universitaria Careggi - S.O.D. Patologia Medica, Florence
- Catharina Ziekenhuis, Eindhoven, Netherlands
- Spain (3):
  - Vall d'Hebron University Hospital, Barcelona
  - Hospital Universitari de Bellvitge, Barcelona
  - Clinica Universidad de Navarra, Pamplona

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- VIZAMYL™: Participants who received a single VIZAMYL™ injection intravenously prior to positron emission tomography (PET) brain imaging, as per the clinical practice.
- All Clinical Readers: Clinical readers had been trained to interpret VIZAMYL™ images using an in-person training programme. They read the Vizamyl images.
Period: Overall Study
Arm/Group | VIZAMYL™ | All Clinical Readers
Started | 209 | 18
Completed | 209 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analysis was performed on all participants that is participants who were enrolled in the study and received a dose of VIZAMYL™ and Clinical readers who read the Vizamyl images.
Groups:
- VIZAMYL™: Participants who received a single VIZAMYL™ injection intravenously prior to PET brain imaging, as per the clinical practice.
- Total: Total of all reporting groups
Arm/Group | VIZAMYL™ | All Clinical Readers | Total
Number analyzed (Participants) | 209 | 18 | 227
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.1 (8.81) | 51.3 (98.4) | NA (NA) — Total age data in any form is unavailable, as it was not planned to calculate data for both arms together. Total Data was not planned and collected.
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 101 | 7 | 108
  Male | 108 | 11 | 119
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 176 | 15 | 191
  Other | 1 | 1 | 2
  Not Reported | 2 | 0 | 2
  Missing | 30 | 2 | 32

OUTCOME MEASURES:

1. Primary Outcome: Accuracy of VIZAMYL™ PET Image Interpretations Made by Clinical Readers
Description: Accuracy was estimated as 100 percent (%) *(number of true positives [TP] + number of true negatives [TN]) / (number of TP + number of TN + number of false positives [FP] + number of false negatives [FN]). The data presented are the point estimates representing percentage of accuracy, with Measure Type "Number" and 95% exact binomial confidence interval. These have been estimated using Clopper-Pearson method.
Time Frame: Up to 1093 days
Population: The efficacy population included participants who had an interpretable image that had an available standard of truth (SOT) classification (expert majority image interpretation).
Measure: Number (95% Confidence Interval); unit: Percentage of image interpretations
Units Other Than Participants: PET image interpretations
Arm/Group | VIZAMYL™
Number analyzed (Participants) | 209
Number analyzed (PET image interpretations) | 209
Percentage of image interpretations | 83.25 [77.49 to 88.05]

2. Primary Outcome: Sensitivity of VIZAMYL™ PET Image Interpretations Made by Clinical Readers
Description: Sensitivity was defined as 100%*number of TP / (number of TP + number of FN). The data presented are the point estimates representing percentage sensitivity, with Measure Type "Number" and 95% exact binomial confidence interval. These have been estimated using Clopper-Pearson method.
Time Frame: Up to 1093 days
Population: The efficacy population included participants who had an interpretable image that had an available SOT classification (expert majority image interpretation).
Measure: Number (95% Confidence Interval); unit: Percentage of image interpretations
Units Other Than Participants: PET image interpretations
Arm/Group | VIZAMYL™
Number analyzed (Participants) | 209
Number analyzed (PET image interpretations) | 209
Percentage of image interpretations | 92.24 [85.78 to 96.39]

3. Primary Outcome: Specificity of VIZAMYL™ PET Image Interpretations Made by Clinical Readers
Description: Specificity was defined as 100%*number of TN / (number of TN + number of FP). The data presented are the point estimates representing the percentage specificity, with Measure Type "Number" and 95% exact binomial confidence interval. These have been estimated using Clopper-Pearson method.
Time Frame: Up to 1093 days
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of image interpretations
Units Other Than Participants: PET image interpretations
Arm/Group | VIZAMYL™
Number analyzed (Participants) | 209
Number analyzed (PET image interpretations) | 209
Percentage of image interpretations | 72.04 [61.78 to 80.86]

4. Primary Outcome: Positive Predictive Value (PPV) of VIZAMYL™ PET Image Interpretations Made by Clinical Readers
Description: The PPV was defined as 100%*number of TP / (number of TP + number of FP). The data presented are the point estimates representing percentage PPV, with Measure Type "Number" and 95% exact binomial confidence interval. These have been estimated using Clopper-Pearson method.
Time Frame: Up to 1093 days
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of image interpretations
Units Other Than Participants: PET image interpretations
Arm/Group | VIZAMYL™
Number analyzed (Participants) | 209
Number analyzed (PET image interpretations) | 209
Percentage of image interpretations | 80.45 [72.68 to 86.81]

5. Primary Outcome: Negative Predictive Value (NPV) of VIZAMYL™ PET Image Interpretations Made by Clinical Readers
Description: The NPV was defined as 100%*number of TN/ (number of TN + number of FN). The data presented are the point estimates representing percentage NPV, with Measure Type "Number" and 95% exact binomial confidence interval. These have been estimated using Clopper-Pearson method.
Time Frame: Up to 1093 days
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of image interpretations
Units Other Than Participants: PET image interpretations
Arm/Group | VIZAMYL™
Number analyzed (Participants) | 209
Number analyzed (PET image interpretations) | 209
Percentage of image interpretations | 88.16 [78.71 to 94.44]

6. Secondary Outcome: Correlation Coefficient Between Clinical Reader Age and Accuracy
Description: Correlation coefficient was used to assess the correlation between clinical reader age and accuracy. A scatterplot of clinical reader accuracy vs. reader age was plotted to check correlation (coefficient) between accuracy and age.
Time Frame: Up to 1093 days
Population: The efficacy clinical reader population consisted of 18 clinical readers who had interpreted the images included from his/her institution and had at least one of their image interpretations classified as TP, TN, FP, or FN through comparison with the SOT (the expert blinded reader majority interpretation).
Measure: Number; unit: Correlation coefficient
Groups:
- VIZAMYL™- Clinical Readers: Participating clinical readers who interpreted the VIZAMYL™ PET images.
Arm/Group | VIZAMYL™- Clinical Readers
Number analyzed (Participants) | 18
Correlation coefficient | -0.2415

7. Secondary Outcome: Number of Participants With Accuracy Less Than (<) 0.9333 or Greater Than Equal to (>=) 0.9333 in Terms of Sex of Clinical Readers
Description: Number of participants with accuracy < 0.9333 or >= 0.9333 in terms of sex of clinical readers were reported.
Time Frame: Up to 1093 days
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | VIZAMYL™- Clinical Readers
Number analyzed (Participants) | 18
Participants
  Accuracy < 0.9333: Male | 6
  Accuracy < 0.9333: Female | 5
  Accuracy >= 0.9333: Male | 5
  Accuracy >= 0.9333: Female | 2
Statistical Analysis 1: Comparison: VIZAMYL™- Clinical Readers; Test type: Other; p = 0.6371, Fisher Exact

8. Secondary Outcome: Number of Participants With Association of Electronic Training (With or Without In-Person Training) With Clinical Reader Accuracy
Description: Number of participants with association of electronic training (with or without In-person training) with clinical reader accuracy were reported.
Time Frame: Up to 1093 days
Population: The efficacy clinical reader population consisted of 18 clinical readers who had interpreted the images included from his/her institution and had at least one of their image interpretations classified as TP, TN, FP, or FN through comparison with the SOT (the expert blinded reader majority interpretation). Here, 'number analyzed' included all clinical readers who were trained or not trained type with clinical reader accuracy.
Measure: Count of Participants; unit: Participants
Arm/Group | VIZAMYL™- Clinical Readers
Number analyzed (Participants) | 18
Participants
  Accuracy >= 0.9333: Trained electronically: number analyzed (Participants) | 7
  Accuracy >= 0.9333: Trained electronically | 2
  Accuracy >= 0.9333: Not Trained electronically: number analyzed (Participants) | 7
  Accuracy >= 0.9333: Not Trained electronically | 5
  Accuracy < 0.9333: Trained electronically: number analyzed (Participants) | 11
  Accuracy < 0.9333: Trained electronically | 8
  Accuracy < 0.9333: Not Trained electronically: number analyzed (Participants) | 11
  Accuracy < 0.9333: Not Trained electronically | 3
Statistical Analysis 1: Comparison: VIZAMYL™- Clinical Readers; Test type: Other; p = 0.1448, Fisher Exact

9. Secondary Outcome: Number of Participants With Association of In-Person Training (With or Without Electronic Training) With Clinical Reader Accuracy
Description: Number of participants with association of In-person training (with or without electronic training) with clinical reader accuracy were reported.
Time Frame: Up to 1093 days
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | VIZAMYL™- Clinical Readers
Number analyzed (Participants) | 18
Participants
  Accuracy >= 0.9333: Trained in person: number analyzed (Participants) | 7
  Accuracy >= 0.9333: Trained in person | 6
  Accuracy >= 0.9333: Not trained in person: number analyzed (Participants) | 7
  Accuracy >= 0.9333: Not trained in person | 1
  Accuracy < 0.9333: Trained in person: number analyzed (Participants) | 11
  Accuracy < 0.9333: Trained in person | 5
  Accuracy < 0.9333: Not trained in person: number analyzed (Participants) | 11
  Accuracy < 0.9333: Not trained in person | 6
Statistical Analysis 1: Comparison: VIZAMYL™- Clinical Readers; Test type: Other; p = 0.1507, Fisher Exact

10. Secondary Outcome: Number of Participants With Association of Training Type With Clinical Reader Accuracy (Excluding Readers Who Took Both Types)
Description: Number of participants with association of training type with clinical reader accuracy (excluding readers who took both types) were reported.
Time Frame: Up to 1093 days
Population: Efficacy clinical reader population. Here 'Overall number of participants analyzed' included all clinical readers who were trained type with clinical reader accuracy and 'number analyzed' signifies who were trained with clinical reader accuracy at specific category.
Measure: Count of Participants; unit: Participants
Arm/Group | VIZAMYL™- Clinical Readers
Number analyzed (Participants) | 15
Participants
  Accuracy >= 0.9333: Trained electronically only: number analyzed (Participants) | 6
  Accuracy >= 0.9333: Trained electronically only | 1
  Accuracy >= 0.9333: Trained in person only: number analyzed (Participants) | 6
  Accuracy >= 0.9333: Trained in person only | 5
  Accuracy < 0.9333: Trained electronically only: number analyzed (Participants) | 9
  Accuracy < 0.9333: Trained electronically only | 6
  Accuracy < 0.9333: Trained in person only: number analyzed (Participants) | 9
  Accuracy < 0.9333: Trained in person only | 3
Statistical Analysis 1: Comparison: VIZAMYL™- Clinical Readers; Test type: Other; p = 0.1189, Fisher Exact

11. Secondary Outcome: Time From Last Training
Description: Time from last training was reported. Number of readers remaining at timepoint was number of readers with accuracy greater than or equal to 0.9333. All readers met this criterion at time 0 hence, data for all clinical reader is reported. All 18 readers were trained in interpretation of Vizamyl images & as part of their training, had their interpretation accuracy tested using 15 test images. To pass test, a reader had to interpret atleast 14 of 15 images correctly. 14 represents 0.9333 of 15, so each reader had to have an accuracy of atleast 0.9333 in order to pass test. Date on which a reader took his/her test is considered to be Time 0. Each reader's accuracy at a later time was assessed in study.
Time Frame: Retrospective data covering up to 8.1 years
Population: as for outcome 6
Measure: Median (Full Range); unit: Years
Arm/Group | VIZAMYL™- Clinical Readers
Number analyzed (Participants) | 18
Years | 3.45 [1.4 to 8.1]

ADVERSE EVENTS:
Time Frame: Up to 1093 days
Description: Analysis was performed on safety population which included participants who were enrolled in the study and received a dose of VIZAMYL™. Adverse event data was not collected from clinical readers as they have not received VIZAMYL™.
Arm/Group | VIZAMYL™
All-Cause Mortality (participants affected / at risk) | 0/209
Serious Adverse Events (participants affected / at risk) | 0/209
Other Adverse Events (participants affected / at risk) | 0/209

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-06-19): https://cdn.clinicaltrials.gov/large-docs/15/NCT04773015/Prot_000.pdf
  • Statistical Analysis Plan (2021-01-06): https://cdn.clinicaltrials.gov/large-docs/15/NCT04773015/SAP_001.pdf